CLINICAL TRIAL: NCT03917082
Title: LA LEAST- Luminal A, Limited Endocrine Adjuvant Systemic Therapy. A Trial of Abbreviated Hormone Therapy for Low Risk Hormone Receptor Positive, HER2 Negative Early Breast Cancer
Brief Title: Limited Adjuvant Endocrine Therapy for Low Risk Breast Cancer
Acronym: LALEAST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); NanoString Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Caroline Lohrisch, Medical Oncologist, Department head, medical oncology Vancouver Centre, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA LEAST
Record Dates: First submitted 2019-03-18; First posted 2019-04-16 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer Female; Hormone Receptor Positive Tumor
Keywords: endocrine therapy
MeSH Terms: interventions — Tamoxifen; Aromatase Inhibitors

STUDY DESIGN:
Intervention Model Description: Single arm phase II study exploring reducing the duration of endocrine therapy from five to two years in low risk population with early breast cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- standard of care endocrine therapy for two years (Experimental): Standard of care adjuvant endocrine therapy for two years. for postmenopausal women, initial therapy will be aromatase inhibitor unless contraindicated, in which case tamoxifen may be used. For premenopausal and perimenopausal women, initial therapy will be tamoxifen unless contraindicated, in which case an lutenizing hormone releasing hormone (LHRH) agonist with / without aromatase inhibitor may be used.
  Interventions: Drug: Tamoxifen Citrate

INTERVENTIONS:
Drug: Tamoxifen Citrate — current standard of care is 5 years endocrine therapy after early breast cancer. Intervention will test if 2 years is adequate for population with low recurrence risk based on genomic tissue based test
  Other Names: aromatase inhibitor

SUMMARY:
Phase II trial of 2 years of standard adjuvant endocrine therapy after low risk hormone receptor positive, HER2 negative, node negative breast cancer in women older than 50 at diagnosis.

The study hypothesis is that reducing adjuvant endocrine therapy from 5 to 2 years in a population with low risk of breast cancer; as determined by histopathologic criteria and confirmed by low risk genomic analysis using Prosigna®; will be safe and acceptable to this population, and will not compromise the expected excellent breast cancer specific outcomes for this population.

DETAILED DESCRIPTION:
Women older than 50 at diagnosis of an invasive breast cancer which is all of: node negative/N0i+; T1 or T2; low or intermediate grade; with strong or intermediate expression of hormone receptors (ER and PR); and HER2 negative, and who have had adequate local therapy for their tumor, are invited to participate in Prosigna® screening. A sample of their excised tumor is sent for Prosigna® testing. This is a validated and widely approved genomic test to assess recurrence risk in hormone receptor positive/HER2 negative, node negative breast tumors. Tumors with a low risk result, defined as Risk of Recurrence (ROR) less than or equal to 40, are then eligible for enrollment on the LA LEAST study of 2 years of endocrine therapy (tamoxifen for pre/perimenopausal women and aromatase inhibitor for postmenopausal women). To mimic real life, there is flexibility to switch to an alternate standard of care endocrine therapy during the two years if intolerable side effects develop. During the two years of therapy, participants are seen every six months and complete periodic quality of life (QOL) questionnaires designed to measure quality of life, mood, side effects, and anxiety/fear of recurrence. Following two years of therapy, participants have annual study visits until year 10, with similar questionnaires at some but not all time points, and assessment of study endpoints. Primary endpoint is the 5 year distant relapse free interval (DRFI), defined as freedom from distant recurrence or breast cancer death at five years. Secondary endpoints include longitudinal QOL comparisons, 10 year breast cancer free interval and 10 year contralateral breast cancer rate. It is anticipated that about 400 individuals will need to be screened to enroll 290 participants with requisite low score. The sample size is based on an expected 5 year DRFI of 96.8%, one sided alpha of 0.05 and a rejection of the alternate hypothesis if the lower boundary of the one sided confidence interval yields an observed DRFI below 95%.

ELIGIBILITY:
Inclusion Criteria: for Prosigna® screening

* Diagnosis of invasive breast cancer which is:

  * Unifocal or multifocal (not multicentric)
  * Unilateral
  * Moderate or strongly hormone receptor positive
  * HER2 negative
  * Ductal grade 1 or 2, or lobular any grade, or pure tubular (any grade) or pure papillary (any grade). If mixed lobular-ductal histology, the ductal component must be grade 1 or 2.
  * Stage pT1N0 (tumor </= 20mm, negative node) or pT2N0 (tumor 21-50mm, node negative) or pT1N0i+ (tumor </=20mm and isolated tumor cells in node[s]) or pT2N0i+ (tumor 21-50mm and isolated tumor cells in node[s]) (see Appendix 2). Tumor size must be sufficient for Prosigna® testing. pNX (nodal status unknown) stage is not eligible.
* Subject must be female
* Subject must be age > 50 years at breast cancer diagnosis
* Subject may be pre, peri, or postmenopausal.
* Subject must have a > 5-year life expectancy based on physician judgement of subject's co-morbid illnesses and age
* Subject must undergo standard of care loco-regional management (sentinel node biopsy and/or axillary dissection; breast conserving surgery or mastectomy; radiation to breast following breast conserving surgery, with radiotherapy details per local institution practice). Surgery will have been no more than 24 weeks prior to endocrine therapy start. Subjects having repeat surgeries after radiation, regardless of indication, should count the date of last surgery that preceded radiation. Subjects may undergo Prosigna® screening prior to completion of radiation.
* The breast surgery will have achieved negative surgical margins. Tumours with positive margins that are not re-resectable are eligible if followed by radiation with a boost (partial mastectomy) or chest wall radiation (mastectomy)
* No (neoadjuvant or adjuvant) chemotherapy given or planned for this breast cancer
* No other non-breast cancer within the last 5 years, except non-melanoma skin cancer, melanoma in situ, cervix carcinoma in situ, and anal carcinoma in situ
* No prior hormone receptor positive invasive breast cancer. Prior contralateral DCIS treated with standard of care local therapy, and prior lobular carcinoma in situ (LCIS) are allowed, provided no endocrine therapy with any of tamoxifen, ovarian suppression, raloxifene, or aromatase inhibitor was given
* Subject will have not have started endocrine therapy prior to enrollment
* Subject has signed a screening informed consent form
* Subject has intent to be adherent to endocrine therapy for two years in the absence of serious toxicity

Inclusion criteria for study enrollment:

* Prosigna® score in the low risk range, defined as an ROR of 40 or lower
* Subject has not yet initiated endocrine therapy
* Subject has signed study informed consent form

Exclusion Criteria:

• Does not meet every inclusion criteria listed above

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer incidence ratio in women vs men is 10:1. Given the sample size of the study, it is unlikely that enrolling men will provide any meaningful data about the impact of limited endocrine therapy for male breast cancer.
Enrollment: 290 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Distant Relapse Free Interval at five years | 5 years after the last patient is enrolled
  freedom from distant recurrence or breast cancer death at 5 years

SECONDARY OUTCOMES:
Ten year breast cancer free interval | ten years after the last patient is enrolled
  freedom from local, regional, distant breast cancer recurrence or death from breast cancer or ipsilateral or contralateral ductal carcinoma in situ or contralateral invasive breast cancer at ten years
Ten year contralateral breast cancer incidence | ten years after the last patient is enrolled
  breast cancer occurring in the contralateral breast, including ductal carcinoma in situ (DCIS) and invasive breast cancer, within ten years of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Lohrisch, MC, Study Chair — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
summary results for participants will be shared in peer review meetings and publications

REFERENCES:
- [Background] Burstein HJ, Temin S, Anderson H, Buchholz TA, Davidson NE, Gelmon KE, Giordano SH, Hudis CA, Rowden D, Solky AJ, Stearns V, Winer EP, Griggs JJ. Adjuvant endocrine therapy for women with hormone receptor-positive breast cancer: american society of clinical oncology clinical practice guideline focused update. J Clin Oncol. 2014 Jul 20;32(21):2255-69. doi: 10.1200/JCO.2013.54.2258. Epub 2014 May 27. PMID 24868023
- [Background] Gnant M, Thomssen C, Harbeck N. St. Gallen/Vienna 2015: A Brief Summary of the Consensus Discussion. Breast Care (Basel). 2015 Apr;10(2):124-30. doi: 10.1159/000430488. PMID 26195941
- [Background] Tamoxifen for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1998 May 16;351(9114):1451-67. PMID 9605801
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Ekholm M, Bendahl PO, Ferno M, Nordenskjold B, Stal O, Ryden L. Two Years of Adjuvant Tamoxifen Provides a Survival Benefit Compared With No Systemic Treatment in Premenopausal Patients With Primary Breast Cancer: Long-Term Follow-Up (> 25 years) of the Phase III SBII:2pre Trial. J Clin Oncol. 2016 Jul 1;34(19):2232-8. doi: 10.1200/JCO.2015.65.6272. Epub 2016 May 9. PMID 27161974
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Cameron DA, Palmer MJ, Pater JL. Randomized trial of letrozole following tamoxifen as extended adjuvant therapy in receptor-positive breast cancer: updated findings from NCIC CTG MA.17. J Natl Cancer Inst. 2005 Sep 7;97(17):1262-71. doi: 10.1093/jnci/dji250. PMID 16145047
- [Background] Davies C, Pan H, Godwin J, Gray R, Arriagada R, Raina V, Abraham M, Medeiros Alencar VH, Badran A, Bonfill X, Bradbury J, Clarke M, Collins R, Davis SR, Delmestri A, Forbes JF, Haddad P, Hou MF, Inbar M, Khaled H, Kielanowska J, Kwan WH, Mathew BS, Mittra I, Muller B, Nicolucci A, Peralta O, Pernas F, Petruzelka L, Pienkowski T, Radhika R, Rajan B, Rubach MT, Tort S, Urrutia G, Valentini M, Wang Y, Peto R; Adjuvant Tamoxifen: Longer Against Shorter (ATLAS) Collaborative Group. Long-term effects of continuing adjuvant tamoxifen to 10 years versus stopping at 5 years after diagnosis of oestrogen receptor-positive breast cancer: ATLAS, a randomised trial. Lancet. 2013 Mar 9;381(9869):805-16. doi: 10.1016/S0140-6736(12)61963-1. PMID 23219286
- [Background] Goss PE, Ingle JN, Pritchard KI, Robert NJ, Muss H, Gralow J, Gelmon K, Whelan T, Strasser-Weippl K, Rubin S, Sturtz K, Wolff AC, Winer E, Hudis C, Stopeck A, Beck JT, Kaur JS, Whelan K, Tu D, Parulekar WR. Extending Aromatase-Inhibitor Adjuvant Therapy to 10 Years. N Engl J Med. 2016 Jul 21;375(3):209-19. doi: 10.1056/NEJMoa1604700. Epub 2016 Jun 5. PMID 27264120
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Aromatase inhibitors versus tamoxifen in early breast cancer: patient-level meta-analysis of the randomised trials. Lancet. 2015 Oct 3;386(10001):1341-1352. doi: 10.1016/S0140-6736(15)61074-1. Epub 2015 Jul 23. PMID 26211827
- [Background] Tjan-Heijnen VCG, van Hellemond IEG, Peer PGM, Swinkels ACP, Smorenburg CH, van der Sangen MJC, Kroep JR, De Graaf H, Honkoop AH, Erdkamp FLG, van den Berkmortel FWPJ, de Boer M, de Roos WK, Linn SC, Imholz ALT, Seynaeve CM; Dutch Breast Cancer Research Group (BOOG) for the DATA Investigators. Extended adjuvant aromatase inhibition after sequential endocrine therapy (DATA): a randomised, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1502-1511. doi: 10.1016/S1470-2045(17)30600-9. Epub 2017 Oct 12. PMID 29031778
- [Background] Love RR, Van Dinh N, Quy TT, Linh ND, Tung ND, Shen TZ, Hade EM, Young GS, Jarjoura D. Survival after adjuvant oophorectomy and tamoxifen in operable breast cancer in premenopausal women. J Clin Oncol. 2008 Jan 10;26(2):253-7. doi: 10.1200/JCO.2007.11.6061. Epub 2007 Dec 17. PMID 18086800
- [Background] Systemic treatment of early breast cancer by hormonal, cytotoxic, or immune therapy. 133 randomised trials involving 31,000 recurrences and 24,000 deaths among 75,000 women. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1992 Jan 11;339(8785):71-85. No abstract available. PMID 1345869
- [Background] Systemic treatment of early breast cancer by hormonal, cytotoxic, or immune therapy. 133 randomised trials involving 31,000 recurrences and 24,000 deaths among 75,000 women. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1992 Jan 4;339(8784):1-15. PMID 1345950
- [Background] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Background] Gnant M, Mlineritsch B, Schippinger W, Luschin-Ebengreuth G, Postlberger S, Menzel C, Jakesz R, Seifert M, Hubalek M, Bjelic-Radisic V, Samonigg H, Tausch C, Eidtmann H, Steger G, Kwasny W, Dubsky P, Fridrik M, Fitzal F, Stierer M, Rucklinger E, Greil R; ABCSG-12 Trial Investigators; Marth C. Endocrine therapy plus zoledronic acid in premenopausal breast cancer. N Engl J Med. 2009 Feb 12;360(7):679-91. doi: 10.1056/NEJMoa0806285. PMID 19213681
- [Background] Gnant M, Mlineritsch B, Stoeger H, Luschin-Ebengreuth G, Knauer M, Moik M, Jakesz R, Seifert M, Taucher S, Bjelic-Radisic V, Balic M, Eidtmann H, Eiermann W, Steger G, Kwasny W, Dubsky P, Selim U, Fitzal F, Hochreiner G, Wette V, Sevelda P, Ploner F, Bartsch R, Fesl C, Greil R; Austrian Breast and Colorectal Cancer Study Group, Vienna, Austria. Zoledronic acid combined with adjuvant endocrine therapy of tamoxifen versus anastrozol plus ovarian function suppression in premenopausal early breast cancer: final analysis of the Austrian Breast and Colorectal Cancer Study Group Trial 12. Ann Oncol. 2015 Feb;26(2):313-20. doi: 10.1093/annonc/mdu544. Epub 2014 Nov 17. PMID 25403582
- [Background] Gnant M, Sestak I, Filipits M, Dowsett M, Balic M, Lopez-Knowles E, Greil R, Dubsky P, Stoeger H, Rudas M, Jakesz R, Ferree S, Cowens JW, Nielsen T, Schaper C, Fesl C, Cuzick J. Identifying clinically relevant prognostic subgroups of postmenopausal women with node-positive hormone receptor-positive early-stage breast cancer treated with endocrine therapy: a combined analysis of ABCSG-8 and ATAC using the PAM50 risk of recurrence score and intrinsic subtype. Ann Oncol. 2015 Aug;26(8):1685-91. doi: 10.1093/annonc/mdv215. Epub 2015 May 1. PMID 25935792
- [Background] Chirgwin JH, Giobbie-Hurder A, Coates AS, Price KN, Ejlertsen B, Debled M, Gelber RD, Goldhirsch A, Smith I, Rabaglio M, Forbes JF, Neven P, Lang I, Colleoni M, Thurlimann B. Treatment Adherence and Its Impact on Disease-Free Survival in the Breast International Group 1-98 Trial of Tamoxifen and Letrozole, Alone and in Sequence. J Clin Oncol. 2016 Jul 20;34(21):2452-9. doi: 10.1200/JCO.2015.63.8619. Epub 2016 May 23. PMID 27217455
- [Background] Baum M, Budzar AU, Cuzick J, Forbes J, Houghton JH, Klijn JG, Sahmoud T; ATAC Trialists' Group. Anastrozole alone or in combination with tamoxifen versus tamoxifen alone for adjuvant treatment of postmenopausal women with early breast cancer: first results of the ATAC randomised trial. Lancet. 2002 Jun 22;359(9324):2131-9. doi: 10.1016/s0140-6736(02)09088-8. PMID 12090977
- [Background] Amir E, Seruga B, Niraula S, Carlsson L, Ocana A. Toxicity of adjuvant endocrine therapy in postmenopausal breast cancer patients: a systematic review and meta-analysis. J Natl Cancer Inst. 2011 Sep 7;103(17):1299-309. doi: 10.1093/jnci/djr242. Epub 2011 Jul 9. PMID 21743022
- [Background] Fontaine C, Meulemans A, Huizing M, Collen C, Kaufman L, De Mey J, Bourgain C, Verfaillie G, Lamote J, Sacre R, Schallier D, Neyns B, Vermorken J, De Greve J. Tolerance of adjuvant letrozole outside of clinical trials. Breast. 2008 Aug;17(4):376-81. doi: 10.1016/j.breast.2008.02.006. Epub 2008 May 2. PMID 18455395
- [Background] Neugut AI, Subar M, Wilde ET, Stratton S, Brouse CH, Hillyer GC, Grann VR, Hershman DL. Association between prescription co-payment amount and compliance with adjuvant hormonal therapy in women with early-stage breast cancer. J Clin Oncol. 2011 Jun 20;29(18):2534-42. doi: 10.1200/JCO.2010.33.3179. Epub 2011 May 23. PMID 21606426
- [Background] Saha P, Regan MM, Pagani O, Francis PA, Walley BA, Ribi K, Bernhard J, Luo W, Gomez HL, Burstein HJ, Parmar V, Torres R, Stewart J, Bellet M, Perello A, Dane F, Moreira A, Vorobiof D, Nottage M, Price KN, Coates AS, Goldhirsch A, Gelber RD, Colleoni M, Fleming GF; SOFT; TEXT Investigators; International Breast Cancer Study Group. Treatment Efficacy, Adherence, and Quality of Life Among Women Younger Than 35 Years in the International Breast Cancer Study Group TEXT and SOFT Adjuvant Endocrine Therapy Trials. J Clin Oncol. 2017 Sep 20;35(27):3113-3122. doi: 10.1200/JCO.2016.72.0946. Epub 2017 Jun 27. PMID 28654365
- [Background] Bernhard J, Luo W, Ribi K, Colleoni M, Burstein HJ, Tondini C, Pinotti G, Spazzapan S, Ruhstaller T, Puglisi F, Pavesi L, Parmar V, Regan MM, Pagani O, Fleming GF, Francis PA, Price KN, Coates AS, Gelber RD, Goldhirsch A, Walley BA. Patient-reported outcomes with adjuvant exemestane versus tamoxifen in premenopausal women with early breast cancer undergoing ovarian suppression (TEXT and SOFT): a combined analysis of two phase 3 randomised trials. Lancet Oncol. 2015 Jul;16(7):848-58. doi: 10.1016/S1470-2045(15)00049-2. Epub 2015 Jun 16. PMID 26092816
- [Background] Ganz PA, Petersen L, Castellon SA, Bower JE, Silverman DH, Cole SW, Irwin MR, Belin TR. Cognitive function after the initiation of adjuvant endocrine therapy in early-stage breast cancer: an observational cohort study. J Clin Oncol. 2014 Nov 1;32(31):3559-67. doi: 10.1200/JCO.2014.56.1662. Epub 2014 Sep 29. PMID 25267747
- [Background] Marino JL, Saunders CM, Emery LI, Green H, Doherty DA, Hickey M. How does adjuvant chemotherapy affect menopausal symptoms, sexual function, and quality of life after breast cancer? Menopause. 2016 Sep;23(9):1000-8. doi: 10.1097/GME.0000000000000664. PMID 27272225
- [Background] Chin SN, Trinkaus M, Simmons C, Flynn C, Dranitsaris G, Bolivar R, Clemons M. Prevalence and severity of urogenital symptoms in postmenopausal women receiving endocrine therapy for breast cancer. Clin Breast Cancer. 2009 May;9(2):108-17. doi: 10.3816/CBC.2009.n.020. PMID 19433392
- [Background] Land SR, Wickerham DL, Costantino JP, Ritter MW, Vogel VG, Lee M, Pajon ER, Wade JL 3rd, Dakhil S, Lockhart JB Jr, Wolmark N, Ganz PA. Patient-reported symptoms and quality of life during treatment with tamoxifen or raloxifene for breast cancer prevention: the NSABP Study of Tamoxifen and Raloxifene (STAR) P-2 trial. JAMA. 2006 Jun 21;295(23):2742-51. doi: 10.1001/jama.295.23.joc60075. Epub 2006 Jun 5. PMID 16754728
- [Background] Henry NL, Banerjee M, Wicha M, Van Poznak C, Smerage JB, Schott AF, Griggs JJ, Hayes DF. Pilot study of duloxetine for treatment of aromatase inhibitor-associated musculoskeletal symptoms. Cancer. 2011 Dec 15;117(24):5469-75. doi: 10.1002/cncr.26230. Epub 2011 Jun 20. PMID 21692065
- [Background] Coleman R, Cameron D, Dodwell D, Bell R, Wilson C, Rathbone E, Keane M, Gil M, Burkinshaw R, Grieve R, Barrett-Lee P, Ritchie D, Liversedge V, Hinsley S, Marshall H; AZURE investigators. Adjuvant zoledronic acid in patients with early breast cancer: final efficacy analysis of the AZURE (BIG 01/04) randomised open-label phase 3 trial. Lancet Oncol. 2014 Aug;15(9):997-1006. doi: 10.1016/S1470-2045(14)70302-X. Epub 2014 Jul 15. PMID 25035292
- [Background] Loprinzi CL, Kugler JW, Sloan JA, Mailliard JA, LaVasseur BI, Barton DL, Novotny PJ, Dakhil SR, Rodger K, Rummans TA, Christensen BJ. Venlafaxine in management of hot flashes in survivors of breast cancer: a randomised controlled trial. Lancet. 2000 Dec 16;356(9247):2059-63. doi: 10.1016/S0140-6736(00)03403-6. PMID 11145492
- [Background] Elston CW, Ellis IO. Pathological prognostic factors in breast cancer. I. The value of histological grade in breast cancer: experience from a large study with long-term follow-up. Histopathology. 1991 Nov;19(5):403-10. doi: 10.1111/j.1365-2559.1991.tb00229.x. PMID 1757079
- [Background] Coombes RC, Powles TJ, Berger U, Wilson P, McClelland RA, Gazet JC, Trott PA, Ford HT. Prediction of endocrine response in breast cancer by immunocytochemical detection of oestrogen receptor in fine-needle aspirates. Lancet. 1987 Sep 26;2(8561):701-3. doi: 10.1016/s0140-6736(87)91071-3. PMID 2888939
- [Background] Sparano JA, Gray RJ, Makower DF, Pritchard KI, Albain KS, Hayes DF, Geyer CE Jr, Dees EC, Goetz MP, Olson JA Jr, Lively T, Badve SS, Saphner TJ, Wagner LI, Whelan TJ, Ellis MJ, Paik S, Wood WC, Ravdin PM, Keane MM, Gomez Moreno HL, Reddy PS, Goggins TF, Mayer IA, Brufsky AM, Toppmeyer DL, Kaklamani VG, Berenberg JL, Abrams J, Sledge GW Jr. Adjuvant Chemotherapy Guided by a 21-Gene Expression Assay in Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):111-121. doi: 10.1056/NEJMoa1804710. Epub 2018 Jun 3. PMID 29860917
- [Background] Paik S, Tang G, Shak S, Kim C, Baker J, Kim W, Cronin M, Baehner FL, Watson D, Bryant J, Costantino JP, Geyer CE Jr, Wickerham DL, Wolmark N. Gene expression and benefit of chemotherapy in women with node-negative, estrogen receptor-positive breast cancer. J Clin Oncol. 2006 Aug 10;24(23):3726-34. doi: 10.1200/JCO.2005.04.7985. Epub 2006 May 23. PMID 16720680
- [Background] Sparano JA, Gray RJ, Makower DF, Pritchard KI, Albain KS, Hayes DF, Geyer CE Jr, Dees EC, Perez EA, Olson JA Jr, Zujewski J, Lively T, Badve SS, Saphner TJ, Wagner LI, Whelan TJ, Ellis MJ, Paik S, Wood WC, Ravdin P, Keane MM, Gomez Moreno HL, Reddy PS, Goggins TF, Mayer IA, Brufsky AM, Toppmeyer DL, Kaklamani VG, Atkins JN, Berenberg JL, Sledge GW. Prospective Validation of a 21-Gene Expression Assay in Breast Cancer. N Engl J Med. 2015 Nov 19;373(21):2005-14. doi: 10.1056/NEJMoa1510764. Epub 2015 Sep 27. PMID 26412349
- [Background] Cardoso F, van't Veer LJ, Bogaerts J, Slaets L, Viale G, Delaloge S, Pierga JY, Brain E, Causeret S, DeLorenzi M, Glas AM, Golfinopoulos V, Goulioti T, Knox S, Matos E, Meulemans B, Neijenhuis PA, Nitz U, Passalacqua R, Ravdin P, Rubio IT, Saghatchian M, Smilde TJ, Sotiriou C, Stork L, Straehle C, Thomas G, Thompson AM, van der Hoeven JM, Vuylsteke P, Bernards R, Tryfonidis K, Rutgers E, Piccart M; MINDACT Investigators. 70-Gene Signature as an Aid to Treatment Decisions in Early-Stage Breast Cancer. N Engl J Med. 2016 Aug 25;375(8):717-29. doi: 10.1056/NEJMoa1602253. PMID 27557300
- [Background] Nielsen TO, Parker JS, Leung S, Voduc D, Ebbert M, Vickery T, Davies SR, Snider J, Stijleman IJ, Reed J, Cheang MC, Mardis ER, Perou CM, Bernard PS, Ellis MJ. A comparison of PAM50 intrinsic subtyping with immunohistochemistry and clinical prognostic factors in tamoxifen-treated estrogen receptor-positive breast cancer. Clin Cancer Res. 2010 Nov 1;16(21):5222-32. doi: 10.1158/1078-0432.CCR-10-1282. Epub 2010 Sep 13. PMID 20837693
- [Background] Dowsett M, Sestak I, Lopez-Knowles E, Sidhu K, Dunbier AK, Cowens JW, Ferree S, Storhoff J, Schaper C, Cuzick J. Comparison of PAM50 risk of recurrence score with oncotype DX and IHC4 for predicting risk of distant recurrence after endocrine therapy. J Clin Oncol. 2013 Aug 1;31(22):2783-90. doi: 10.1200/JCO.2012.46.1558. Epub 2013 Jul 1. PMID 23816962
- [Background] Kelly CM, Bernard PS, Krishnamurthy S, Wang B, Ebbert MT, Bastien RR, Boucher KM, Young E, Iwamoto T, Pusztai L. Agreement in risk prediction between the 21-gene recurrence score assay (Oncotype DX(R)) and the PAM50 breast cancer intrinsic Classifier in early-stage estrogen receptor-positive breast cancer. Oncologist. 2012;17(4):492-8. doi: 10.1634/theoncologist.2012-0007. Epub 2012 Mar 14. PMID 22418568
- [Background] Wallden B, Storhoff J, Nielsen T, Dowidar N, Schaper C, Ferree S, Liu S, Leung S, Geiss G, Snider J, Vickery T, Davies SR, Mardis ER, Gnant M, Sestak I, Ellis MJ, Perou CM, Bernard PS, Parker JS. Development and verification of the PAM50-based Prosigna breast cancer gene signature assay. BMC Med Genomics. 2015 Aug 22;8:54. doi: 10.1186/s12920-015-0129-6. PMID 26297356
- [Background] Laenkholm AV, Jensen MB, Eriksen JO, Rasmussen BB, Knoop AS, Buckingham W, Ferree S, Schaper C, Nielsen TO, Haffner T, Kibol T, Moller Talman ML, Bak Jylling AM, Tabor TP, Ejlertsen B. PAM50 Risk of Recurrence Score Predicts 10-Year Distant Recurrence in a Comprehensive Danish Cohort of Postmenopausal Women Allocated to 5 Years of Endocrine Therapy for Hormone Receptor-Positive Early Breast Cancer. J Clin Oncol. 2018 Mar 10;36(8):735-740. doi: 10.1200/JCO.2017.74.6586. Epub 2018 Jan 25. PMID 29369732
- [Background] Cella D, Fallowfield LJ. Recognition and management of treatment-related side effects for breast cancer patients receiving adjuvant endocrine therapy. Breast Cancer Res Treat. 2008 Jan;107(2):167-80. doi: 10.1007/s10549-007-9548-1. Epub 2007 Sep 18. PMID 17876703
- [Background] Cossetti RJ, Tyldesley SK, Speers CH, Zheng Y, Gelmon KA. Comparison of breast cancer recurrence and outcome patterns between patients treated from 1986 to 1992 and from 2004 to 2008. J Clin Oncol. 2015 Jan 1;33(1):65-73. doi: 10.1200/JCO.2014.57.2461. Epub 2014 Nov 24. PMID 25422485
- [Background] Viani GA, Afonso SL, Stefano EJ, De Fendi LI, Soares FV. Adjuvant trastuzumab in the treatment of her-2-positive early breast cancer: a meta-analysis of published randomized trials. BMC Cancer. 2007 Aug 8;7:153. doi: 10.1186/1471-2407-7-153. PMID 17686164
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res. 1997 Jan;42(1):17-41. doi: 10.1016/s0022-3999(96)00216-4. PMID 9055211
- [Background] Hagen KB, Aas T, Kvaloy JT, Eriksen HR, Soiland H, Lind R. Fatigue, anxiety and depression overrule the role of oncological treatment in predicting self-reported health complaints in women with breast cancer compared to healthy controls. Breast. 2016 Aug;28:100-6. doi: 10.1016/j.breast.2016.05.005. Epub 2016 Jun 2. PMID 27262826
- [Background] Taira N, Shimozuma K, Shiroiwa T, Ohsumi S, Kuroi K, Saji S, Saito M, Iha S, Watanabe T, Katsumata N. Associations among baseline variables, treatment-related factors and health-related quality of life 2 years after breast cancer surgery. Breast Cancer Res Treat. 2011 Aug;128(3):735-47. doi: 10.1007/s10549-011-1631-y. Epub 2011 Jun 17. PMID 21681445
- [Background] Gotay CC, Pagano IS. Assessment of Survivor Concerns (ASC): a newly proposed brief questionnaire. Health Qual Life Outcomes. 2007 Mar 13;5:15. doi: 10.1186/1477-7525-5-15. PMID 17352831
- [Background] Radtke JV, Terhorst L, Cohen SM. The Menopause-Specific Quality of Life Questionnaire: psychometric evaluation among breast cancer survivors. Menopause. 2011 Mar;18(3):289-95. doi: 10.1097/gme.0b013e3181ef975a. PMID 20881889
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630